CLINICAL TRIAL: NCT01181609
Title: An Open-label Study of Avastin in Combination With Chemotherapy Regimens as Second-line Treatment in Patients With Metastatic Colon or Rectal Cancer
Brief Title: A Study of Avastin (Bevacizumab) Combined With Chemotherapy in Patients With Metastatic Cancer of the Colon or Rectum
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML18559
Record Dates: First submitted 2010-07-30; First posted 2010-08-13 (Estimated); Results first posted 2014-07-28 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: bevacizumab [Avastin]

INTERVENTIONS:
Drug: bevacizumab [Avastin] — 5 mg/kg every 2 weeks or 7.5 mg/kg every 3 weeks according to the chemotherapy regimen

SUMMARY:
This study will assess the efficacy and safety of intravenous Avastin in combination with chemotherapy regimens as second-line treatment of metastatic cancer of the colon or rectum. The anticipated time of study treatment is until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic colon or rectal cancer, progressing or relapsing after first-line treatment;
* Women of childbearing potential must use adequate contraception up to at least 6 months after the last dose of bevacizumab.

Exclusion Criteria:

* Patients with metastatic colon or rectal cancer scheduled for a first-line systemic treatment;
* Untreated brain metastases, spinal cord compression or primary brain tumours;
* Pregnant or lactating women;
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study start;
* Treatment with any investigational drug, or participation in another investigational study, within 30 days prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2005-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (16):
- France (16):
  - Angers
  - Besançon
  - Boulogne-Billancourt
  - Colmar
  - Dijon
  - La Roche-sur-Yon
  - Marseille
  - Montpellier
  - Neuilly-sur-Seine
  - Nice
  - Paris
  - Pierre-Bénite
  - Reims
  - Saint-Cloud
  - Saint-Herblain
  - Toulouse

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab + Chemotherapy: Participants received bevacizumab 2.5 milligrams per kilogram (mg/kg) intravenously (IV) per week, either as 5 mg/kg on Day 1 of a 2-week cycle or as 7.5 mg/kg on Day 1 of a 3-week cycle and was dependent on the chemotherapy regimen used. The choice of chemotherapy regimen was left to the discretion of the investigator per standard of care at the study site. Cycle was repeated until disease progression or withdrawal of participant.
Period: Overall Study
Arm/Group | Bevacizumab + Chemotherapy
Started | 54
Completed | 1
Not Completed | 53
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1
Not completed — Death | 50

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: included participants who received at least 1 dose of treatment.
Groups:
- Bevacizumab + Chemotherapy: Participants received bevacizumab 2.5 mg/kg IV per week, either as 5 mg/kg on Day 1 of a 2-week cycle or as 7.5 mg/kg on Day 1 of a 3-week cycle and was dependent on the chemotherapy regimen used. The choice of chemotherapy regimen was left to the discretion of the investigator per standard of care at the study site. Cycle was repeated until disease progression or withdrawal of participant.
Arm/Group | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 35

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Overall Disease Control (ODC)
Description: ODC was defined as the percentage of participants with measurable disease at baseline who on assessment achieved complete response (CR), partial response (PR), or stable disease (SD) according to Response Evaluation Criteria in Solid Tumors (RECIST). CR defined as disappearance of all target lesions, non-target lesions, and normalization of tumor marker level. PR was defined as greater than or equal to (≥) 30 percent (%) decrease under baseline of the sum of the longest diameter (LD) of all target lesions. SD defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum LD since start of treatment. CR and PR were confirmed no less than 4 weeks after the criteria for response were met.
Time Frame: Baseline, after every other cycle to disease progression or death (Maximum of 52.5 months follow-up)
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 53
percentage of participants | 87 [77 to 97]

2. Secondary Outcome: Percentage of Participants Achieving a Best Overall Response of CR or PR
Description: Percentage of participants achieving CR or PR as defined by RECIST criteria. CR defined as disappearance of all target lesions, non-target lesions, and normalization of tumor marker level. PR was defined as ≥30% decrease under baseline of the sum of the LD of all target lesions. CR and PR were confirmed no less than 4 weeks after the criteria for response were met.
Time Frame: Baseline, every cycle to progression or death (Maximum of 52.5 months follow-up)
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 53
percentage of participants | 32 [19 to 46]

3. Secondary Outcome: Progression-Free Survival (PFS) - Percentage of Participants With an Event
Description: PFS was defined as the time from start of study treatment to investigator assessed disease progression, or death due to any cause, whichever comes first. Progression was based on tumor assessments made by the investigators according to RECIST.
Time Frame: Baseline, every cycle to progression or death (Maximum of 52.5 months follow-up)
Population: ITT
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 53
percentage of participants | 98

4. Secondary Outcome: PFS - Time to Event
Description: PFS was defined as the time from start of study treatment to investigator assessed disease progression, or death due to any cause, whichever comes first. Progression was based on tumor assessments made by the investigators according to RECIST. Median PFS was estimed using the Kaplan-Meier method.
Time Frame: Baseline, every cycle to progression or death (Maximum of 52.5 months follow-up)
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 53
months | 6.5 [5.8 to 7.8]

5. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the time in months from the day of CR or PR was first noted to the day of progression of disease, death or last follow-up. Median duraiton of response is estimated sing the Kaplan-Meier method.
Time Frame: Baseline, every cycle until progression or death (Maximum of 52.5 months follow-up)
Population: ITT population; only participants with a response (CR or PR) were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 17
months | 6 [4.8 to 7.5]

6. Secondary Outcome: Duration of Overall Disease Control
Description: ODC duration was defined as the time in months, from when measurement criteria were first met for CR, PR, or SD (whichever status was recorded first) until the first date when progressive disease or the death from any cause was documented. Data were censored for participants who were lost to follow-up, discontinued prematurely without progression/death, or who reached the end of study without progression. Median ODC was estimated using the Kaplan-Meier method.
Time Frame: Baseline, every cycle until progression or death. (Maximum of 52.5 months follow-up)
Population: ITT population; only participants with an ODC response (CR, PR, or SD) were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 46
months | 6.7 [5.2 to 7.1]

7. Secondary Outcome: Overall Survival (OS) - Percentage of Participants With an Event
Description: Overall survival was defined as the time from start of study treatment to death from any cause.
Time Frame: Baseline, every cycle to progression or death (Maximum of 52.5 months follow-up)
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 53
percentage of participants | 93.0

8. Secondary Outcome: OS - Time to Event
Description: OS was defined as the time from start of study treatment to death from any cause. Median OS was estimated using the Kaplan-Meier method.
Time Frame: Baseline, every cycle to progression or death. (Maximum of 52.5 months follow-up)
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 53
months | 19.3 (14,2) [14.2 to 25.1]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were reported from the data of first study-drug administration until 28 days after the last study-drug administration.
Description: All participants who received at least 1 dose of study treatment were included in the safety analysis population.
Arm/Group | Bevacizumab + Chemotherapy
Serious Adverse Events (participants affected / at risk) | 9/53
Other Adverse Events (participants affected / at risk) | 52/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Chemotherapy (N=53)
Abdominal pain (Gastrointestinal disorders) | 3
Hyperthermia (General disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Gastroenteritis (Infections and infestations) | 1
Renal failure (Renal and urinary disorders) | 1
Renal pain (Renal and urinary disorders) | 1
Inguinal hernia repair (Surgical and medical procedures) | 1
Radiofrequency ablation (Surgical and medical procedures) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Colonoscopy (Surgical and medical procedures) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Cholinergic syndrome (Psychiatric disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Chemotherapy (N=53)
Nausea (Gastrointestinal disorders) | 35
Diarrhea (Gastrointestinal disorders) | 32
Vomiting (Gastrointestinal disorders) | 25
Abdominal pain (Gastrointestinal disorders) | 13
Constipation (Gastrointestinal disorders) | 12
Abdominal pain upper (Gastrointestinal disorders) | 8
Aphthous stomatitis (Gastrointestinal disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 5
Toothache (Gastrointestinal disorders) | 4
Haemorrhoids (Gastrointestinal disorders) | 3
Asthenia (General disorders) | 32
Mucosal inflammation (General disorders) | 18
Fatigue (General disorders) | 6
Pyrexia (General disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 18
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 6
Paresthesia (Nervous system disorders) | 13
Headache (Nervous system disorders) | 8
Neuropathy (Nervous system disorders) | 5
Dizziness (Nervous system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 16
Anemia (Blood and lymphatic system disorders) | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Gastroenteritis (Infections and infestations) | 5
Rhinitis (Infections and infestations) | 4
Nasopharyngitis (Infections and infestations) | 3
Anorexia (Metabolism and nutrition disorders) | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Weight decreased (Investigations) | 4
Anxiety (Psychiatric disorders) | 5
Eye disorder (Eye disorders) | 8
Surgical and medical procedures (Surgical and medical procedures) | 5
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 4
Vascular disorders (Vascular disorders) | 3
Hepatobiliary disorders (Hepatobiliary disorders) | 3
Renal and urinary disorders (Renal and urinary disorders) | 3
Hypertension (Vascular disorders) | 22
Bleeding/hemorrhage (all epistaxis) (Respiratory, thoracic and mediastinal disorders) | 29
Gastro-intestinal perforation (Gastrointestinal disorders) | 0
Wound healing complication (Injury, poisoning and procedural complications) | 1
Proteinuria (Renal and urinary disorders) | 6
Thromboembolism (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request the Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.